CLINICAL TRIAL: NCT02436668
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Phase 3 Study of the Bruton's Tyrosine Kinase Inhibitor Ibrutinib in Combination With Nab-paclitaxel and Gemcitabine Versus Placebo in Combination With Nab-paclitaxel and Gemcitabine, in the First Line Treatment of Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Study of Ibrutinib vs Placebo, in Combination With Nab-paclitaxel and Gemcitabine, in the First Line Treatment of Patients With Metastatic Pancreatic Adenocarcinoma (RESOLVE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCYC-1137-CA
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — ibrutinib; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibrutinib (Active Comparator): Ibrutinib daily in combination with:
  Nab-paclitaxel and gemcitabine
  Interventions: Drug: Ibrutinib; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Placebo (Placebo Comparator): Placebo daily in combination with:
  Nab-paclitaxel and gemcitabine
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Ibrutinib
  Other Names: IMBRUVICA®
  Arms: Ibrutinib
Drug: Gemcitabine
Drug: Nab-paclitaxel

SUMMARY:
This is a phase 3 study to evaluate the efficacy of ibrutinib in combination with nab-paclitaxel and gemcitabine for the first line treatment of patients with metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma.
2. Stage IV disease diagnosed within 6 weeks of randomization
3. Adequate hematologic function:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Hemoglobin ≥9 g/dL
4. Adequate hepatic and renal function defined as:

   * AST and/or ALT ≤5.0 x upper limit of normal (ULN) if liver metastases, or ≤3 x ULN without liver metastases
   * Alkaline phosphatase <3.0 x ULN or ≤5.0 x ULN if liver or bone metastases present
   * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin, such as hemolysis)
   * Estimated Creatinine Clearance ≥30 mL/min
5. PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN
6. KPS ≥70.
7. Eastern Cooperative Oncology Group (ECOG) 0-1

Exclusion Criteria:

1. Prior therapies: BTK inhibitor, radiotherapy, radiotherapy in the adjuvant setting, or cytotoxic chemotherapy for primary disease of pancreatic adenocarcinoma.
2. Neuroendocrine (carcinoid, islet cell) or acinar pancreatic carcinoma
3. Known brain or leptomeningeal disease (CT or MRI scan of the brain required only in case of clinical suspicion of central nervous system involvement).
4. Major surgery within 4 weeks of first dose of study drug.
5. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
6. Treatment with a strong cytochrome P450 (CYP) 3A inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2015-05; Primary Completion 2018-10 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Cole, MD, Study Director — Pharmacyclics LLC.
Locations (86):
- United States (28):
  - Oncology Specialties, PC; Clearview Cancer Institute, Huntsville, Alabama
  - Arizona Center for Cancer Care, Avondale, Arizona
  - St. Mary's Medical Center, Daly City, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology/Oncology Assoc., Norwich, Connecticut
  - Bethesda Memorial Hospital, Boynton Beach, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Ingalls Memorial Hospital Cancer Research Center, Harvey, Illinois
  - Joliet Oncology-Hematology Associates, LTD, Joliet, Illinois
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Berkshire Hematology Oncology Services at Berkshire Medical Center Cancer and Infusion Center, Pittsfield, Massachusetts
  - Saint Joseph Mercy Health System, Chelsea, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Nebraska Medicine - Peggy D. Cowdery Patient Care Center, Omaha, Nebraska
  - The Presbyterian Hospital, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Penn State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Scott & White Memorial Hospital, Temple, Texas
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
- Belgium (5):
  - ULB Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Gilly
  - UZ Leuven, Leuven
  - C. H. U. Sart Tilman, Liège
- France (11):
  - Centre Antoine Lacassagne, Nice, Alpes Maritimes
  - Centre Paul Strauss, Strasbourg, Bas Rhin
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - Groupe Hospitalier Saint André - Hôpital Saint André, Bordeaux, Gironde
  - CHU de Toulouse - Hôpital Rangueil, Toulouse, Haute Garonne
  - Hôpital Nord Franche Comté, Doubs, Montbeliard
  - Hôpital Saint-Antoine, Paris, Paris
  - CHU Poitiers - Hôpital la Milétrie, Poitiers, Vienne
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Germany (7):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Gemeinschaftspraxis Haematologie und Onkologie, Dresden, Saxony-Anhalt
  - Onkologische Schwerpunktpraxis Kurfuerstendamm, Berlin
- Italy (10):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Ancona
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Ospedale San Raffaele, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- South Korea (8):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (10):
  - ICO l´Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Specialist, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (7):
  - Derriford Hospital, Plymouth, Devon
  - Broomfield Hospital, Chelmsford, Essex
  - The Christie, Manchester, Greater Manchester
  - Southampton General Hospital, Southampton, Hampshire
  - The Clatterbridge Cancer Centre, Liverpool, Merseyside
  - Royal Marsden Hospital, Sutton, Surrey
  - Royal Free Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 75 centers in the United States (US), European Union, and South Korea. The first subject enrolled 08 May 2015 and the last was enrolled on April 19, 2018.
Pre-assignment Details: There was a safety run-in of 6 patients; subsequently, 430 total patients were enrolled. Eligible subjects were required to have a confirmed diagnosis of Stage IV pancreatic adenocarcinoma within 6 weeks of randomization evaluable per RECIST 1.1 criteria with at least 1 measurable metastatic lesion. Key exclusion criteria included any previous cytotoxic chemotherapy for primary disease of pancreatic adenocarcinoma.
Groups:
- Placebo+Gemcitabine+Nab-Paclitaxel: Placebo daily in combination with:
  Nab-paclitaxel and gemcitabine
  Nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 were administered on Days 1, 8, and 15 of each 28-day cycle, each as a 30- to 40-minute intravenous infusion
- Ibrutinib+Gemcitabine+Nab-paclitaxel: Ibrutinib daily in combination with:
  Nab-paclitaxel and gemcitabine
  Ibrutinib was administered orally once daily at a starting dose of 560 mg.
  Nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 were administered on Days 1, 8, and 15 of each 28-day cycle, each as a 30- to 40-minute intravenous infusion.
Period: Overall Study
Arm/Group | Placebo+Gemcitabine+Nab-Paclitaxel | Ibrutinib+Gemcitabine+Nab-paclitaxel
Started | 213 | 211
Completed | 212 | 207
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Pbo+n-P/G: Placebo daily in combination with:
  Nab-paclitaxel and gemcitabine
  Nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 were administered on Days 1, 8, and 15 of each 28-day cycle, each as a 30- to 40-minute intravenous infusion.
- Ibr+n-P/G: Ibrutinib daily in combination with:
  Nab-paclitaxel and gemcitabine
  Ibrutinib- orally once daily at a starting dose of 560 mg.
  Nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 were administered on Days 1, 8, and 15 of each 28-day cycle, each as a 30- to 40-minute intravenous infusion
- Total: Total of all reporting groups
Arm/Group | Pbo+n-P/G | Ibr+n-P/G | Total
Number analyzed (Participants) | 213 | 211 | 424
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 119 | 118 | 237
  >=65 years | 94 | 93 | 187
Age, Continuous [Median (Full Range); unit: Years] | 64.0 [32 to 85] | 64.0 [32 to 82] | 64.0 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 97 | 189
  Male | 121 | 114 | 235
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 18
  Not Hispanic or Latino | 197 | 198 | 395
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 59 | 53 | 112
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 142 | 146 | 288
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization until disease progression per RECIST 1.1 criteria assessed by investigator, or death from any cause, whichever occurs first.
Time Frame: Results at an overall median follow-up of 24.87 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib+Gemcitabine+Nab-paclitaxel | Placebo+Gemcitabine+Nab-Paclitaxel
Number analyzed (Participants) | 211 | 213
Months | 5.32 [3.75 to 5.49] | 6.01 [5.45 to 7.16]
Statistical Analysis 1: Comparison: Ibrutinib+Gemcitabine+Nab-paclitaxel vs Placebo+Gemcitabine+Nab-Paclitaxel; The treatment effect was tested with an stratified log rank test. Hazard ratio is estimated using Cox regression model stratified by the three randomization stratification factors [KPS (70 80 vs. 90-100), liver metastasis (present vs. absent), and age (≤65 vs. >65)] and with treatment as the only covariate; Test type: Superiority; p < 0.0001, Log Rank — P-value is from log-rank test stratified by the three randomization stratification factors [KPS (70-80 vs. 90-100), liver metastasis (present vs. absent), and age (≤65 vs. >65)]; Hazard Ratio (HR) = 1.525, 95% CI 2-sided [1.241 to 1.873]

2. Primary Outcome: Overall Survival (OS)
Description: OS, is defined as the time from date of randomization until date of death from any cause.
Time Frame: Results at an overall median follow-up of 24.87 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib+Gemcitabine+Nab-paclitaxel | Placebo+Gemcitabine+Nab-Paclitaxel
Number analyzed (Participants) | 211 | 213
Months | 9.69 [8.57 to 10.41] | 10.78 [8.94 to 11.66]
Statistical Analysis 1: Comparison: Ibrutinib+Gemcitabine+Nab-paclitaxel vs Placebo+Gemcitabine+Nab-Paclitaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — P-value is based on log-rank test stratified by the three randomization stratification factors [KPS (70-80 vs. 90-100), liver metastasis (present vs. absent), and age (≤65 vs. >65)]; p = 0.3225, Log Rank; Hazard Ratio (HR) = 1.109, 95% CI 2-sided [0.903 to 1.363]

3. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Ibrutinib and Nab-paclitaxel and Gemcitabine Versus Placebo in Combination With Nab-paclitaxel and Gemcitabine.
Description: This is a measure of percentage of subjects with Treatment Emergent Adverse Events Grade 3 or above collected Up to 30 days after the last participating subject discontinues study drug.
Time Frame: Results at an overall median follow-up of 24.87 months
Population: The safety population included 420 subjects and was used for the analyses of all safety endpoints and included all subjects in the ITT population who received at least 1 dose of study drug (ibrutinib, placebo, nab-paclitaxel, or gemcitabine). The data sets analyzed are summarized in the following table.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+Gemcitabine+Nab-Paclitaxel | Ibrutinib+Gemcitabine+Nab-paclitaxel
Number analyzed (Participants) | 212 | 208
percentage of participants
  Subjects with any TEAE >= Grade 3 | 86.8 | 85.6
  Subjects with ibrutinib/pbo-related TEAE >=Grade 3 | 55.7 | 54.3

4. Secondary Outcome: Overall Response Rate
Description: ORR is defined as the percentage of subjects who achieve a complete response or partial response, based on investigator assessment according to RECIST 1.1.
Time Frame: Results at an overall median follow-up of 24.87 months
Measure: Number (95% Confidence Interval); unit: percentage of Patients
Arm/Group | Placebo+Gemcitabine+Nab-Paclitaxel | Ibrutinib+Gemcitabine+Nab-paclitaxel
Number analyzed (Participants) | 213 | 211
percentage of Patients | 42.3 [35.5 to 49.2] | 29.5 [23.3 to 36]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Nab-Paclitaxel vs Ibrutinib+Gemcitabine+Nab-paclitaxel; For rate ratio, numerator is Ibr+Gem/Abr arm and denominator is Pbo + Gem/Abr arm. P-value for rate ratio is based on Cochran-Mantel-Haenszel (CMH) test adjusted for the three randomization stratification factors. Two-sided 95% confidence interval for rate ratio is based on Mantel-Haenszel method; Test type: Superiority; p = 0.0058, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.695, 95% CI 2-sided [0.535 to 0.903]

5. Secondary Outcome: Clinical Benefit Response
Description: Subject achieved a ≥50% reduction in pain intensity (Memorial Pain Assessment Card [MPAC]) or analgesic consumption, or a 20-point or greater improvement in KPS for a period of at least 4 consecutive weeks, without showing any sustained worsening in other parameters.
  OR Subject was stable on all of the aforementioned parameters, and showed a marked, sustained weight gain (≥7% increase maintained for ≥4 weeks) not due to fluid accumulation (Burris 1997).
Time Frame: Results at an overall median follow-up of 24.87 months
Population: Clinical benefit response rate was not analyzed due to incomplete data for the analgesic use. Data for subjects who "Achieved a >=50% reduction in pain intensity", "20-point or greater improvement in KPS (>=4 consecutive weeks)", "Sustained weight gain (>=7% increase maintained for >=4 weeks) not due to fluid accumulation"are reported.
Measure: Number; unit: percentage of patients
Groups:
- Ibrutinib+Gemcitabine+Nab-paclitaxel: Ibrutinib daily in combination with:
  Nab-paclitaxel and gemcitabine Ibrutinib was administered orally once daily at a starting dose of 560 mg. Nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 were administered on Days 1, 8, and 15 of each 28-day cycle, each as a 30- to 40-minute intravenous infusion.
  I
Arm/Group | Placebo+Gemcitabine+Nab-Paclitaxel | Ibrutinib+Gemcitabine+Nab-paclitaxel
Number analyzed (Participants) | 213 | 211
percentage of patients
  Achieved a >=50% reduction in pain intensity | 25.8 | 27.5
  >=20-pt improvement in KPS (>=4 consecutive weeks) | 1.4 | 0
  Sustained weight gain (>=7% maintained >4 weeks | 11.7 | 5.7

6. Secondary Outcome: Carbohydrate Antigen 19-9 (CA19-9) Response
Description: The CA19-9 response rate is defined as the percentage of subjects with a decline of 20%, 90%, and other thresholds considered clinically meaningful, from baseline. This is a percentage of patients with > or = 60% reduction from baseline.
Time Frame: Results at an overall median follow-up of 24.87 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Placebo+Gemcitabine+Nab-Paclitaxel | Ibrutinib+Gemcitabine+Nab-paclitaxel
Number analyzed (Participants) | 213 | 211
percentage of patients | 62.9 [56.0 to 69.4] | 53.6 [46.6 to 60.4]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Nab-Paclitaxel vs Ibrutinib+Gemcitabine+Nab-paclitaxel; For rate ratio, numerator is Ibr+Gem/Abr arm and denominator is Pbo+Gem/Abr arm. P-value for rate ratio is based on Cochran-Mantel-Haenszel (CMH) test adjusted for the three randomization stratification factors. Two-sided 95% confidence interval for rate ratio is based on Mantel-Haenszel method; Test type: Superiority; p = 0.0488, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.850, 95% CI 2-sided [0.722 to 1.0] — This 0.85 (0.722 to 1.0) with CI is referring to risk ratio not proportional/percentage of patients

7. Secondary Outcome: Patient-reported Outcome (PRO) by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30).
Description: Unit is the month: TUDD1 - the time between random & 1st occurrence of a decrease in QLQ-C30 score ≥10 pts w/o improvement in QoL score of ≥10 points or any further QoL data due to deterioration. The proportion of subjects who met the "responder" criteria prior to subsequent anticancer therapy initiation. Response defined as achievement of a ≥50% reduction in MPAC visual analog scale which measures pain intensity or analgesic consumption, or a ≥20-point improvement from baseline in KPS sustained for a period of ≥ 4 consecutive weeks without showing any sustained worsening from baseline in any of the other parameters OR Subject stable on all parameters (pain and KPS), & showed a marked, sustained weight gain (≥7% increase from baseline maintained for ≥4 weeks) not due to fluid accumulation.
Time Frame: Results at an overall median follow-up of 24.87 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+Gemcitabine+Nab-Paclitaxel | Ibrutinib+Gemcitabine+Nab-paclitaxel
Number analyzed (Participants) | 213 | 211
months | 6.14 [4.86 to 8.21] | 4.21 [2.86 to 5.82]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Nab-Paclitaxel vs Ibrutinib+Gemcitabine+Nab-paclitaxel; [1] Hazard ratio is based on a Cox proportional hazards model stratified by the three randomization stratification factors for time until definitive deterioration (TUDD1), a hazard ratio < 1 favors Ibr + Gem/Abr. TUDD1 is defined as the time interval between randomization and the first occurrence of a decrease in score by >= 10 points without any further improvement in score by >= 10 points or any further available QoL data due to dropout after deterioration; Test type: Superiority; p = 0.0782, Log Rank — P-value is from log-rank test stratified by the three randomization stratification factors; Hazard Ratio (HR) = 1.265, 95% CI 2-sided [0.975 to 1.642]

8. Secondary Outcome: Rate of Venous Thromboembolic Events (VTE)
Description: The VTE rate is defined as percentage of subjects with Venous thromboembolic events (SMQ) per investigator assessment.
Time Frame: Results at an overall median follow-up of 24.87 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo+Gemcitabine+Nab-Paclitaxel | Ibrutinib+Gemcitabine+Nab-paclitaxel
Number analyzed (Participants) | 213 | 211
Percentage of Participants | 10.8 [7.0 to 15.8] | 8.1 [4.8 to 12.6]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Nab-Paclitaxel vs Ibrutinib+Gemcitabine+Nab-paclitaxel; For rate of VTEs, denominator is number of subjects in the Intent-to-Treat population and numerator is number of Intent-to-Treat subjects with at least one VTE observed any time on study. Confidence interval for rate of VTEs is based on Clopper-Pearson method. [1] P value is based on Chi-square test; Test type: Superiority; p = 0.3343, Chi-squared

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug
Description: There were 4 patient that was randomized but off study without any treatment. This patient had received baseline assessments and included in all efficacy analysis but was excluded from safety population, i.e. not at risk for AE assessment.
Groups:
- Placebo (Plus Nab-paclitaxel and Gemcitabine): Placebo daily in combination with:
  Nab-paclitaxel and gemcitabine
  Nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 were administered on Days 1, 8, and 15 of each 28-day cycle, each as a 30- to 40-minute intravenous infusion
- Ibrutinib (Plus Nab-paclitaxel and Gemcitabine): Ibrutinib 560 mg (4 x 140 mg capsules) (or placebo) was administered orally once daily beginning on Day 1 of Cycle 1 of the treatment phase, with the first dose of ibrutinib given no more than 72 hours after randomization
  Nab-paclitaxel 125 mg/m2 and gemcitabine 1000 mg/m2 were administered on Days 1, 8, and 15 of each 28-day cycle, each as a 30- to 40-minute intravenous infusion
Arm/Group | Placebo (Plus Nab-paclitaxel and Gemcitabine) | Ibrutinib (Plus Nab-paclitaxel and Gemcitabine)
All-Cause Mortality (participants affected / at risk) | 188/212 | 189/208
Serious Adverse Events (participants affected / at risk) | 127/212 | 112/208
Other Adverse Events (participants affected / at risk) | 211/212 | 208/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Plus Nab-paclitaxel and Gemcitabine) (N=212) | Ibrutinib (Plus Nab-paclitaxel and Gemcitabine) (N=208)
Anaemia (Blood and lymphatic system disorders) | 9 (13) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 6 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6) | 4 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (4)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 14 (17)
Vomiting (Gastrointestinal disorders) | 6 (6) | 5 (9)
Abdominal pain (Gastrointestinal disorders) | 11 (12) | 4 (7)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 4 (6)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 17 (20) | 13 (16)
Asthenia (General disorders) | 7 (7) | 6 (8)
General physical health deterioration (General disorders) | 5 (6) | 4 (5)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 4 (6) | 9 (14)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 4 (4) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (11) | 13 (14)
Cellulitis (Infections and infestations) | 1 (1) | 4 (4)
Infection (Infections and infestations) | 1 (1) | 4 (4)
Liver abscess (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Bacteraemia (Infections and infestations) | 0 (0) | 3 (3)
Escherichia sepsis (Infections and infestations) | 1 (2) | 3 (3)
Biliary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 3 (3) | 1 (1)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 3 (4) | 1 (2)
Vascular device infection (Infections and infestations) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 4 (5) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (4) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Enzyme abnormality (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 6 (7)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (8) | 5 (6)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (3)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (4)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Wernicke's encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Plus Nab-paclitaxel and Gemcitabine) (N=212) | Ibrutinib (Plus Nab-paclitaxel and Gemcitabine) (N=208)
Anaemia (Blood and lymphatic system disorders) | 95 (309) | 90 (289)
Thrombocytopenia (Blood and lymphatic system disorders) | 55 (208) | 75 (221)
Neutropenia (Blood and lymphatic system disorders) | 84 (328) | 68 (139)
Leukopenia (Blood and lymphatic system disorders) | 18 (61) | 15 (19)
Vision blurred (Eye disorders) | 15 (18) | 17 (20)
Diarrhoea (Gastrointestinal disorders) | 109 (240) | 147 (357)
Nausea (Gastrointestinal disorders) | 107 (242) | 116 (228)
Vomiting (Gastrointestinal disorders) | 86 (184) | 85 (169)
Constipation (Gastrointestinal disorders) | 78 (96) | 68 (91)
Abdominal pain (Gastrointestinal disorders) | 67 (99) | 63 (94)
Abdominal pain upper (Gastrointestinal disorders) | 27 (40) | 38 (64)
Stomatitis (Gastrointestinal disorders) | 21 (28) | 36 (50)
Dyspepsia (Gastrointestinal disorders) | 21 (26) | 34 (38)
Ascites (Gastrointestinal disorders) | 25 (35) | 21 (30)
Abdominal distension (Gastrointestinal disorders) | 13 (13) | 13 (15)
Asthenia (General disorders) | 93 (283) | 100 (311)
Pyrexia (General disorders) | 82 (181) | 85 (150)
Fatigue (General disorders) | 65 (170) | 78 (149)
Oedema peripheral (General disorders) | 77 (143) | 60 (97)
Mucosal inflammation (General disorders) | 19 (29) | 24 (36)
Chills (General disorders) | 15 (21) | 21 (24)
Urinary tract infection (Infections and infestations) | 16 (25) | 16 (23)
Nasopharyngitis (Infections and infestations) | 15 (17) | 7 (10)
Weight decreased (Investigations) | 21 (33) | 14 (19)
Platelet count decreased (Investigations) | 17 (61) | 13 (26)
Alanine aminotransferase increased (Investigations) | 25 (42) | 12 (16)
Neutrophil count decreased (Investigations) | 19 (48) | 11 (19)
Aspartate aminotransferase increased (Investigations) | 18 (34) | 8 (12)
Decreased appetite (Metabolism and nutrition disorders) | 76 (129) | 85 (135)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (32) | 25 (37)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16 (28) | 17 (24)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (16) | 11 (14)
Dehydration (Metabolism and nutrition disorders) | 12 (14) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 35 (58) | 28 (36)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (38) | 25 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (30) | 17 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (31) | 17 (24)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 11 (13)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 (15) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 63 (153) | 69 (171)
Paraesthesia (Nervous system disorders) | 20 (42) | 27 (79)
Headache (Nervous system disorders) | 20 (24) | 21 (25)
Dizziness (Nervous system disorders) | 20 (22) | 20 (22)
Dysgeusia (Nervous system disorders) | 26 (33) | 19 (24)
Neuropathy peripheral (Nervous system disorders) | 14 (28) | 15 (33)
Neurotoxicity (Nervous system disorders) | 18 (47) | 14 (40)
Peripheral motor neuropathy (Nervous system disorders) | 11 (23) | 13 (30)
Insomnia (Psychiatric disorders) | 34 (36) | 20 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (27) | 36 (41)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 43 (64) | 25 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (47) | 15 (19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 (22) | 9 (14)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 87 (119) | 90 (130)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 (42) | 23 (28)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7) | 14 (16)
Rash erythematous (Skin and subcutaneous tissue disorders) | 15 (21) | 12 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (36) | 8 (8)
Hypotension (Vascular disorders) | 13 (15) | 12 (15)
Hypertension (Vascular disorders) | 13 (34) | 11 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Institution/Investigator will not publish without Sponsor prior review and approval
2. Institution/Investigator will not publish until the earlier of (i) results of study are submitted for publication (ii) notification that submission of the multicenter results are no longer planned (iii) 18 months after study termination.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT02436668/SAP_000.pdf
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02436668/Prot_001.pdf